CLINICAL TRIAL: NCT00698321
Title: Liberia School-Based HIV/STD Prevention Program
Brief Title: A School-Based HIV/STD Prevention Program to Reduce Risky Sexual Behaviors Among Adolescents in Liberia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen B. Kennedy, Principal Investigator, Pacific Institute for Research and Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21MH082666 (NIH); R21MH082666 (NIH); DAHBR 9A-ASPA
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: HIV/STD Prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participating schools will deliver HIV/STD prevention modules.
  Interventions: Behavioral: HIV/STD prevention curriculum
- 2 (Active Comparator): Participating schools will deliver general health promotion modules.
  Interventions: Behavioral: General health promotion curriculum

INTERVENTIONS:
Behavioral: HIV/STD prevention curriculum — The curriculum will include eight 1-hour HIV prevention modules administered weekly for 8 weeks. The modules will educate youth about risky sexual behaviors and will provide them with knowledge and skills necessary to reduce their risk of STDs, HIV, and pregnancy by abstaining from sex or using condoms if they choose to have sex. The curriculum is based on cognitive behavioral theories, focus groups, and the researchers' experience working with youth.
  Other Names: Making Proud Choices!
  Arms: 1
Behavioral: General health promotion curriculum — The curriculum will include eight 1-hour general health modules administered weekly for 8 weeks. The curriculum will focus on teaching students healthful behaviors, including eating habits, physical activity, dental hygiene, and avoidance of cigarette smoking and substance abuse.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a school-based HIV/sexually transmitted disease prevention program in reducing sexual risk behaviors of youth attending school in Liberia.

DETAILED DESCRIPTION:
Currently, more than 60 million people have been diagnosed with HIV/AIDS worldwide. It is estimated that about two-thirds of all HIV infections are among people in Africa. The African country of Liberia, in particular, is experiencing an increase in HIV/sexually transmitted disease (STD) infections and is in need of improved HIV/STD-related prevention programs. With the majority of the new infections occurring among people who are between 15 and 29 years old, new HIV/STD prevention programs are needed to educate youth about proper condom use and risks associated with sexual behaviors. Previous research has suggested that behavioral interventions can reduce adolescents' sexual behaviors that are tied to risk of acquiring STDs. The evidenced-based HIV prevention program, Making Proud Choices, is an intervention originally designed for community settings in the United States, but is currently being adapted in schools of certain sub-Saharan African countries. Adapting this community-based curriculum to school-based settings and cultural contexts within Liberia may be effective in reducing risky sexual behaviors in Liberian adolescents. This study will compare the effectiveness of a school-based HIV/STD prevention program that draws on the curriculum of Making Proud Choices versus a general health promotion program in reducing sexual risk behaviors of youth attending school in Liberia.

Participation in this study will involve two phases. Phase 1 will last 8 months and will be used to adapt the community-based curriculum of Making Proud Choices to school-based settings and contexts within Liberia. Data to guide the integration and cultural adaptation of the curriculum will be collected from school administrators, students, health educators, and community-based organizations through focus groups, group discussions, and interviews.

Phase 2 will last about 12 months and will include junior high schools in Liberia. Participating schools will be assigned randomly to provide the adapted HIV prevention curriculum or a general health promotion curriculum. Before starting course modules, students receiving either curriculum will complete questionnaires about their risk-associated sexual behaviors and knowledge about condom use and abstinence. Both curriculums will include eight 1-hour modules delivered weekly over 8 weeks. The HIV prevention curriculum will focus on increasing knowledge about preventing HIV, STDs, and pregnancy; improving condom use skills; increasing confidence in the ability to negotiate safer sex and to use condoms correctly; and lowering the incidence of sexual-risk behavior. The general health promotion curriculum will focus on teaching students healthful behaviors, including eating habits, physical activity, dental hygiene, and avoidance of cigarette smoking and substance abuse. All participants will repeat the initial questionnaires immediately after completing the curriculum and 3, 6, and 9 months after the curriculum ends.

ELIGIBILITY:
Inclusion Criteria:

* A 6th or 7th grader attending school in Liberia

Exclusion Criteria:

* Not enrolled in the study schools

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 866 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Frequency of unprotected sex | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B. Kennedy, MD, MPH, Principal Investigator — Pacific Institute for Research and Evaluation
Locations (1):
- University of Liberia, Monrovia, Montserrado County, Liberia